CLINICAL TRIAL: NCT05644210
Title: The Clinical Efficacy and Safety of Telitacicept Followed With Rituximab Therapy on APS Secondary to SLE ，a Multicentre Observational Study
Brief Title: Telitacicept Followed With Rituximab Therapy on APS Secondary to SLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Shu, Principal Investigator, Qilu Hospital of Shandong University
Other Study IDs: Bioagents in APS QiluH
Record Dates: First submitted 2022-11-17; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Antiphospholipid Syndrome
Keywords: Telitacicept; Rituximab
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — telitacicept; Rituximab; Aspirin; Agouti Signaling Protein; Warfarin; Hydroxychloroquine; Prednisone; prednylidene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood, saliva and stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RTX+TA group: Screening stage：Patients received 200mg of rituximab intravenously at week 0 and week 2.
  Follow-up period：Telitacicept 160mg once a week for 24 weeks Basic treatment： Hydroxychloroquine、Prednisone、Warfarin、Aspirin
  Interventions: Drug: Telitacicept; Drug: Rituximab; Drug: Aspirin; Drug: Warfarin; Drug: Hydroxychloroquine; Drug: Prednisone
- RTX group: Screening stage：Patients received 200mg of rituximab intravenously at week 0 and week 2.
  Follow-up period Basic treatment：Hydroxychloroquine、Prednisone、Warfarin、Aspirin
  Interventions: Drug: Rituximab; Drug: Aspirin; Drug: Warfarin; Drug: Hydroxychloroquine; Drug: Prednisone

INTERVENTIONS:
Drug: Telitacicept — 160mg once a week for 24 weeks
  Other Names: TA
  Groups: RTX+TA group
Drug: Rituximab — Patients received 200mg of rituximab intravenously at week 0 and week 2.
  Other Names: RTX
Drug: Aspirin — 50-100mg, po, once per day (Qd) prescribed if needed and adjusted due to patient response
  Other Names: Asp
Drug: Warfarin — Warfarin should be used in patients with arterial thrombosis, and rivaroxaban should be replaced if the patient cannot reach the standard or cannot tolerate it
  Other Names: WF
Drug: Hydroxychloroquine — 200mg, po, twice per day (Bid) prescribed，if tolerated by the patient， the dose should remain constant during the observation period
  Other Names: HCQ
Drug: Prednisone — 5-30mg, po, once per day(Qd) prescribed if needed and adjusted due to patient response
  Other Names: Pred

SUMMARY:
The aim of this study was to observe the clinical efficacy and safety of rituximab (RTX) combination with telitacicept (TA) in patients of systemic lupus erythematosus secondary antiphospholipid syndrome (APS).

DETAILED DESCRIPTION:
In this multicenter, prospective, observational study, 80 patients with SLE Secondary APS patients were enrolled. RTX alone or its continuation with TA was observed for 24weeks，and extended for another 24 weeks. At week 12, the RTX group could be converted to the combination group. The primary end point was the response rate of total antiphospholipid antibody (aPL) at week 12. The secondary end points included the decline rate and value of aPL antibody, aGAPSS score, remission degree of specific clinical indicators, changes in SLE disease activity in SAPS group, and drug safety at week 12 and week 24.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients who meet 2006 Sapporo classification criteria of APS or 2020 nonstandard APS performance；

  2.Patients who meet 1997 or 2019 SLE classification criteria ;

  3.Positive LA /ACL/ aβ2GPI ,on two or more occasions, at least 12 weeks apart;

  4.with at least one extra-criteria manifestations of APS, including thrombocytopenia, hemolytic anemia, nephropathy, valve heart disease ,skin ulcer and arterial or deep vein thrombosis;

  5.Maintain a stable base treatment regimen for at least 4 weeks before screening; Basic treatment includes anticoagulants/antiplatelet agents, glucocorticoids, and hydroxychloroquine;

  6.No response, intolerance or dependence on glucocorticoids and immunosuppressants;

  7.Patients who had previously used beliumab or Telitacicept could be enrolled in the study after 12 weeks of discontinuation;

  8.Age ≥18 years;

  9.Signed Informed consent.

Exclusion Criteria:

* 1.Patients with other causes of thrombocytopenia, hemolytic anemia, valvular heart disease, kidney disease and skin ulcer symptoms were excluded, such as drugs, infections, blood system diseases, genetic metabolic diseases, etc;

  2.Severe cardiovascular diseases, kidney, liver and other important organ injuries, serious blood and endocrine system lesions (aplastic anemia, hyperthyroidism crisis, etc.) were excluded; A history of active malignancy (within 5 years) was excluded and chemoradiotherapy was performed; Patients with organ or bone marrow transplantation in the past year were excluded. Exclusion of mentally ill persons;

  3.A history of allergy to the relevant test drug;

  4.Patients had recently received a live vaccine or planned to use any live vaccine during the study;

  5.Ongoing pregnancy;

  6.Patients who were participants in clinical trials of other immunosuppressive agents/biologics within 24 weeks;

  7.Other conditions that the investigator considers would make the candidate unsuitable for the study;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Meet the diagnostic criteria of SLE and related symptoms of secondary APS;
  2. Positive LA /ACL/ aβ2GPI ,on two or more occasions, at least 12 weeks apart;
  3. One or more of the following related clinical symptoms:
  1. Refractory/recurrent thrombocytopenia;
  2. Autoimmune hemolytic anemia;
  3. Heart valve disease;
  4. Renal involvement;
  5. Skin ulcer;
  6. arterial or deep vein thrombosis;
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who achieved response(complete response and partial response) in aPL profiles | Week 12
  For the lupus anticoagulant (LAC) test, we defined complete response (CR) as a negative test result and no response(NR) as a positive test result； For the anticardiolipin antibody (aCL)/anti-β2 glycoprotein I (anti-β2GPI)enzyme-linked immunosorbent assay,CR was defined as a titer of<the 95th percentile, partial response (PR) was defined as a titer of 95th -99th , and NR was defined as a titer of >the 99th percentile.

SECONDARY OUTCOMES:
The proportion of patients who achieved response(complete response and partial response) in aPL profiles | Week 24,48
  For the lupus anticoagulant (LAC) test, we defined complete response (CR) as a negative test result and no response(NR) as a positive test result； For the anticardiolipin antibody (aCL)/anti-β2 glycoprotein I (anti-β2GPI)enzyme-linked immunosorbent assay,CR was defined as a titer of<the 95th percentile, partial response (PR) was defined as a titer of 95th -99th , and NR was defined as a titer of >the 99th percentile.
The change of aPL titer | week 12 , 24,48
  titer change of lupus anticoagulant, anticardiolipin antibody and anti-β2 glycoprotein-I antibody
The changes of the positive number of 7 aPL indicators | week 12, 24,48
  Change in the number of antibody positives.
The change of clinical efficacy in subgroups with different symptoms | Before the screening,baseline and week 12,24,48
  Thrombocytopenia, haemolytic anemia, nephropathy, heart valve lesions, skin changes (livedo reticularis, leg ulcers)
The change of aGAPSS score | Before the screening,baseline and week 12,24,48
  The aGAPSS was calculated by adding the points corresponding to the risk factors: three for hyperlipidemia, one for arterial hypertension, five for positive anticardiolipin antibodies, four for positive anti-β2 glycoprotein-I antibodies and four for positive lupus anticoagulant test.
The change of Damage Index for Antiphospholipid Syndrome (DIAPS) | Before the screening and week 12,24,48
  The score is obtained by adding the output rating for each domain. The instrument demonstrated content, criterion, and construct validity being a precise tool to quantify organ damage in APS.
The change of Physician Global Assessment (PGA) score . | Before the screening,baseline and week 12,24,48
  PGA is a physician-reported visual analogue scale that provides an overall meas- ure of the subject's current disease activity,the PGA is a visual analog scale scored from 0 to 3. A score of 1 corresponds to mild lupus disease activity. A score of 2 correlates with moderate disease activity and a score of 3 with severe disease activity;
The change of Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2k) Score | Before the screening,baseline and week 12,24,48
  The SLEDAI-2K is an established, validated SLE activity index. It is based on the presence of 24 features in 9 organ systems and measures disease activity in SLE patients in the previous 10 days.
The percentage of patients with Lupus Low Disease Activity State (LLDAS) | Before the screening,baseline and week 12,24,48
  LLDAS is defined as: (1) SLE Disease Activity Index (SLEDAI)-2K ≤4, with no activity in major organ systems (renal, central nervous system (CNS), cardiopulmonary, vasculitis, fever) and no haemolytic anaemia or gastrointestinal activity; (2) no new lupus disease activity compared with the previous assessment; (3) a Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA)-SLEDAI physician global assessment (scale 0-3) ≤1; (4) a current prednisolone (or equivalent) dose ≤7.5 mg daily; and (5) well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents.
Glucocorticoid (GC) dose and reduction rate | Before the screening,baseline and week 4,12,24,48
  The proportion of patients who received the GC dose at each time point

OTHER OUTCOMES:
The number of participants experiencing adverse events | Before the screening,baseline and week 4,12,24,48
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiaoyun, Dr., Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China